CLINICAL TRIAL: NCT03862053
Title: A Phase 4 Study to Assess the Clinical Efficacy and Safety of Manuka Eye Drops for Treatment of Allergy
Brief Title: Manuka Eye Droops for Treatment of Allergy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough time to complete trial;covid
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCOPTIMEL-2019
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Allergic Conjunctivitis
Keywords: ocular allergy; allergy; manuka honey; anti-inflammatory
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: randomized, double-blind placebo controlled
Who Masked: Participant, Investigator
Masking Description: medications will be covered by blank labels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Manuka honey eyedrops (Active Comparator): optimel manuka eyedrops 10 ml used as directed in a CAC (Conjunctival allergen challenge) study
  Interventions: Drug: Manuka honey
- Normal saline 0.9% eyedrops (Placebo Comparator): sterile normal saline eyedrops used as directed in a CAC (conjunctival allergen challenge) study
  Interventions: Drug: Manuka honey

INTERVENTIONS:
Drug: Manuka honey — manuka eyedrops applied to the ocular surface
  Other Names: optimel eyedrops

SUMMARY:
Manuka honey eye drops are used for dry eyes and blepharitis. Manuka honey has been proven to be useful for eczema, atopic dermatitis, wound healing, anti-bacterial, anti-parasitic and anti-inflammatory actions.

DETAILED DESCRIPTION:
Ocular allergy is a condition that can affect a patient's quality of life. Symptoms of ocular allergy include but are not limited to red, itchy, swollen, foreign body sensation, watery, puffy or blurry eyes. irritation, redness, burning, foreign body sensation, dryness, pain and blurry vision. In many cases, ocular allergic conjunctivitis are due to seasonal allergens like pollen, mold or indoor allergens such as pet dander or dust mites.

Ocular allergy can be treated by avoidance of known allergens, reduction of allergens by use of HEPA filters, cleaning linens, etc, topical decongestants, over the counter and prescription topical non-steroidals, topical or oral antihistamines, mast cell stabilizers or topical or oral steroids.

Manuka honey is produced by bees that are associated with the flowers of the Manuka plant (Leptospermum scoparium) that grows in New Zealand. Manuka honey is different from other honeys because it has been shown to the more potent due to its higher methylglyoxal concentration.

Manuka honey has been used for its anti-oxidant, anti-bacteral and anti-inflammatory properties. It has been shown to be useful in healing eczematous skin lesions. This study will attempt to demonstrate topical anti-allergy use for ocular allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read, understand and sign and informed consent.
2. Provision of signed and dated informed consent form and HIPPA authorization.
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged 10-85 years.
5. Positive bilateral CAC reaction (> or = to 2 units itching and > or = to 2 units redness in two of three vessel beds) within 10 minutes of instillation of the last allergen titration at visit 1 and a similarly positive bilateral CAC reaction at two or more time points at visit 2.
6. Normal eyelid anatomy
7. BCVA of 20/100 or better in each eye and IOP 5-22 mmHg in both eyes.
8. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of study drug administration
9. Are postmenopausal (no menstrual cycle for at least one year prior to Visit 1) or have undergone bilateral tubal ligation, hysterectomy, hysterectomy with uni- or bilateral oophorectomy, or bilateral oophorectomy.
10. Willingness to avoid the use of disallowed medications and contact lenses for the duration of the clinical trial.

    -

Exclusion Criteria:

1. Have a known hypersensitivity or contraindication to the investigational product or their components.
2. Unwilling to attend study visits.
3. Active ocular disease or significant illness (clinically significant blepharitis, uncontrolled cardiovascular disease, narrow-angle glaucoma) that could affect their safety or the parameters of the study.
4. Contact lens use within the week prior to screening
5. Unwilling to discontinue contact lens use for the duration of the study
6. Pregnancy or lactation
7. Ocular surgery or eyelid surgery within 6 months prior to screening.
8. Subjects must be unwilling to abstain from eyelash growth products containing prostaglandins for the duration of the trial.
9. Subjects must not have had penetrating intraocular surgery, refractive surgery or corneal transplantation, eyelid surgery within 6 months prior to Visit 1.
10. Febrile illness within one week.
11. Treatment with another investigational drug or other intervention within one month.
12. Subjects with a history of herpetic keratitis.
13. Have serious or severe disease or uncontrolled medical condition that in the judgement of the investigator could confound study assessments or limit compliance.
14. Use of new prescription eyedrop within 30 days of screening
15. Change in systemic medication within 30 days of screening
16. Anticipated relocation or extensive travel outside the study site that may preclude compliance with follow up visits over the study period
17. Did not meet CAC requirements at both Visits 1 and 2.

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Estimated)

PRIMARY OUTCOMES:
Subject-assessed ocular itching | 7 weeks
  on a scale from 0-100 where 0 =no itching and 100=maximal itching subtracted scores measured for placebo treatments at visits 3B, 4 and 5
Investigator-assessed conjunctival hyperemia in both eyes at each visit | 7 weeks
  on a scale from 0-100 where 0=no hyperemia and 100=maximal hyperemia subtracted scores from placebo treatments at visits 3B, 4 and 5

SECONDARY OUTCOMES:
investigator-assessed ciliary hyperemia | 7 weeks
  on a scale from 0-100 where 0=no hyperemia and 100=maximal hyperemia subtracted scores from placebo treatments at visits 3B, 4 and 5
investigator assessed episcleral hyperemia | 7 weeks
  on a scale from 0-100 where 0=no hyperemia and 100=maximal hyperemia subtracted scores from placebo treatments at visits 3B, 4 and 5
investigator-assessed chemosis | 7 weeks
  on a scale from 0-100 where 0=no hyperemia and 100=maximal hyperemia subtracted scores from placebo treatments at visits 3B, 4 and 5

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Toyos Clinic, Germantown, Tennessee
  - Toyos Clinic, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
If requested, data records without identifying patient information could be shared